CLINICAL TRIAL: NCT05268939
Title: A Multicenter Study Conducted to Evaluate the Performance of the LumiraDx SARS-CoV-2 & FLU A/B Test, and LumiraDx SARS-CoV-2 & RSV Test at Point of Care Testing Sites
Brief Title: Performance Evaluation of the LumiraDx SARS-CoV-2 & FLU A/B and SARS-CoV-2 & RSV Tests for Aid in the Assessment of COVID-19
Acronym: INSPIRE-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LumiraDx UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-CLIN-PROT-00034
Record Dates: First submitted 2022-03-03; First posted 2022-03-07 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: COVID-19; Influenza A; Influenza Type B; RSV Infection
MeSH Terms: conditions — COVID-19; Respiratory Syncytial Virus Infections

STUDY DESIGN:
Intervention Model Description: Performance Evaluation study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Nasal Swab (Experimental): Nasal swab from subjects with signs and symptoms of COVID-19 and/or Influenza and/or RSV-like illness
  Interventions: Diagnostic Test: LumiraDx SARS-CoV-2 & Flu A/B test; Diagnostic Test: LumiraDx SARS-CoV-2 & RSV test
- Nasopharyngeal Swab (Experimental): Nasopharyngeal swab from subjects with signs and symptoms of COVID-19 and/or Influenza and/or RSV-like illness
  Interventions: Diagnostic Test: LumiraDx SARS-CoV-2 & Flu A/B test; Diagnostic Test: LumiraDx SARS-CoV-2 & RSV test

INTERVENTIONS:
Diagnostic Test: LumiraDx SARS-CoV-2 & Flu A/B test — Swab Samples for Diagnostic test
Diagnostic Test: LumiraDx SARS-CoV-2 & RSV test — Swab Samples for Diagnostic test

SUMMARY:
A Multicenter Study Conducted to Evaluate the Performance of the LumiraDx SARS-CoV-2 & FLU A/B Test, and LumiraDx SARS-CoV-2 & RSV Test at Point of Care Testing Sites. Subjects presenting with symptoms suggestive of COVID-19 and/or Influenza and/or RSV will be consented and asked to donate swab sample(s) for testing in the device(s) under evaluation.

DETAILED DESCRIPTION:
Approximately one-thousand (1000) subjects will be enrolled in this study. Patients presenting to their health care professionals, drive through testing sites or research centers and meet the inclusion/exclusion criteria will be enrolled in the study.

A subject's participation in this study will consist of a single visit. Following completion of the informed consent process and a review of Inclusion/Exclusion criteria to determine eligibility, each subject will receive a unique study identification number.

The potential subject will be asked to provide relevant medical history information (i.e., regarding their influenza/RSV and or COVID-19-like symptoms), which will be evaluated against all inclusion and exclusion criteria depending in their cohort. A subject's SARS-CoV-2 vaccination status will also be collected including the doses, dates of vaccination and brand.

Specimens will be obtained from each subject enrolled using standard collection methods.

The objectives of this study are to:

* Evaluate the performance of the LumiraDx SARS-CoV-2 & Flu A/B Test in detecting SARS-CoV-2 and/ or influenza A or B in nasal and nasopharyngeal swabs from patients with signs and symptoms of COVID-19 or influenza as compared with an FDA EUA authorized or 510(k) comparative method.
* Evaluate the performance of the LumiraDx SARS-CoV-2 & RSV Test in detecting SARS-CoV-2 and/ or RSV in nasal and nasopharyngeal swabs from patients with signs and symptoms of COVID-19 or RSV as compared with an FDA EUA authorized or 510(k) comparative method.
* Evaluate the point of care usability of the LumiraDx SARS-CoV-2 & Flu A/B Test and LumiraDx SARS-CoV-2 & RSV Test.

ELIGIBILITY:
Inclusion Criteria:

1. Preliminary assessment of the subject by the Investigator/designee should be suggestive of COVID-19 and /or influenza and/or RSV at the time of the study visit.
2. The subject must present in one of the following two cohorts:

   Covid Cohort:

   Preliminary assessment of the subject by the Investigator/designee should be suggestive of COVID-19 at the time of the study visit. The subject must present as symptomatic, meaning they have exhibited one or more of the following signs and symptoms for eligibility: fever, cough, shortness of breath, difficulty breathing, muscle pain, headache, sore throat, chills, repeated shaking with chills, new loss of taste or smell, congestion or runny nose, diarrhea, nausea or vomiting. The onset of these symptoms will be recorded and will be in the last twelve (12) days.

   or The subject must have presented with respiratory symptoms and a documented positive SARS-CoV-2 PCR or antigen test in the past forty-eight (48) hours.

   Influenza/RSV Cohort:

   The subject must have a fever of 100.0 °F or greater with the onset of the fever being within the past three (3) days and/or present at the time of the visit. Fever can be reported or taken at time of visit. Subjects must report having a fever, but a quantitative reported measurement is not necessary for inclusion. In addition to the fever, the subject must have two (2) or more of the following signs and symptoms for eligibility: cough, shortness of breath, difficulty breathing, muscle pain, joint pain, headache, chills, repeated shaking with chills, congestion or runny nose, diarrhea, nausea, vomiting, sneezing, sore throat, wheezing, fatigue, weakness and/or malaise or anorexia. The onset of these symptoms will be recorded and will be in the last four (4) days. OR The subject must have presented with respiratory symptoms and a documented positive Flu or RSV test in the past forty-eight (48) hours.
3. Written informed consent must be obtained prior to study enrollment. A subject who is a legal adult must be willing to give written informed consent and must agree to comply with study procedures. The Legal Guardian or Legal Authorized Representative of a subject who is under the age of consent must give written informed consent and agree to comply with study procedures. Active assent should be obtained from children of appropriate intellectual age (as defined by the IRB)

Exclusion Criteria:

1. The subject underwent a nasal wash/aspirate as part of standard of care testing during this study visit.
2. Subjects undergoing treatment currently and/or within the past fourteen (14 days of the study visit with an inhaled influenza vaccine (FluMist®) or with antiviral medication, which may include but is not limited to Amantadine (Symmetrel®), Rimantadine (Flumadine®), Zanamivir (Relenza®), Oseltamivir (Tamiflu®), or Baloxavir Marboxil (Xofluza™)
3. Subjects undergoing treatment currently and/or within the past thirty (30) days of the study with prescription medication to treat novel Coronavirus SARS-CoV-2 infection, which may include but is not limited to Remdesivir (Veklury) or receiving convalescent plasma therapy for SARS-CoV-2;
4. The subject is undergoing treatment currently or had undergone within the past fourteen (14) days of the study visit with RSV-related medication which may include but is not limited to Ribavirin (Virazole), RSV-IGIV (RespiGam) or palivizumab (Synagis).
5. The subject is currently receiving or has received within the past thirty (30) days of the study visit an experimental biologic, drug, or device including either treatment or therapy.
6. The subject has previously participated in this research study (CS-1262-01).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Performance evaluation by health care professionals | 4 months
  Evaluate the performance of the LumiraDx Tests in detecting and differentiating SARS-CoV-2, influenza A, influenza B and/or RSV in fresh nasal or nasopharyngeal swab specimens from patients with signs and symptoms of COVID-19, Influenza and/or RSV-like illness. Performance will be evaluated by use of statistical analysis techniques to assess sensitivity (true positive rate), specificity (true negative rate), Negative and Positive Percent Agreement (NPA, PPA) of the LumiraDx test results versus an FDA-approved method where a result of 100% sensitivity, specificity, NPA or PPA would equate to complete agreement with the reference method and 0% would equate to no agreement.
Point of Care usability | 4 months
  Evaluate the point of care usability of the LumiraDx SARS-CoV-2 & Flu A/B Test and LumiraDx SARS-CoV-2 & RSV Tests. Usability will be assessed by means of a user questionnaire to be completed by naive users following their first test of the devices using standard Pack Leaflet and Quick Reference Instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Ramin Farsad, Principal Investigator — Diagnamics, Inc; Sherri Casey, Principal Investigator — Benchmark Research; Justin Wilson, Principal Investigator — Cullman Clinical Trials; Miguel Perez, Principal Investigator — Excellence Medical and Research; Mary Imig, Principal Investigator — Koch Family Medicine; Marisela Gonzalez, Principal Investigator — Marisela Gonzalez, MD, PA; Lawrence Gervasi, Principal Investigator — Clinical Research Solutions; Rogelio Machuca, Principal Investigator — Machuca Foundation
Locations (8):
- United States (8):
  - Cullman Clinical Trials, Cullman, Alabama
  - Diagnamics, Inc, Encinitas, California
  - Marisela Gonzalez, MD, PA, Miami, Florida
  - Excellence Medical and Research, Miami Gardens, Florida
  - Koch Family Medicine, Morton, Illinois
  - Benchmark Research, Covington, Louisiana
  - Machuca Foundation, Las Vegas, Nevada
  - Clinical Research Solutions, Middleburg Heights, Ohio

IPD SHARING:
Plan to Share IPD: No